CLINICAL TRIAL: NCT03977454
Title: Periarticular Injection Versus Peripheral Nerve Block in Total Hip Arthroplasty: a Single Center Randomized Controlled Trail (RCT) Study
Brief Title: Periarticular Injection Versus Peripheral Nerve Block in Total Hip Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000025198
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Results first posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-08

CONDITIONS: Hip Arthropathy
MeSH Terms: interventions — Nerve Block; Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 patients will receive nerve block per standard of care (Experimental): Nerve blocks (QLB/LFCNB) to be placed preoperatively with dexamethasone sodium phosphate (DEX) and methylprednisolone acetate (MPA), per standard of care of anesthesia block service.
  1. QLB: 40ml 0.2% ropivacaine with 5 mg DEX/ 40 mg MPA; and
  2. LFCNB: 20ml 0.2% ropivacaine with 5 mg DEX/ 40 mg MPA Preoperatively, Group 1 patients will receive nerve block per standard of care as stated above. Intraoperatively, Group 1 will NOT receive PAI.
  Interventions: Procedure: Nerve Block; Drug: Ropivacaine
- Group 2 will NOT receive any nerve blocks. (Active Comparator): Intraoperatively, the surgeon will perform PAI with exactly the same medication as group 1, ie, 60 ml 0.2% ropivacaine and 10 mg DEX/ 80 mg MPA, per standard of care of Surgeon.
  Interventions: Procedure: Periarticular Injection (PAI); Drug: Ropivacaine; Drug: Dex

INTERVENTIONS:
Procedure: Nerve Block — Nerve blocks (QLB/LFCNB) to be placed preoperatively with DEX/MPA, per standard of care of anesthesia block service.
  1. QLB: 40ml 0.2% ropivacaine with 5 mg DEX/ 40 mg MPA
  2. LFCNB: 20ml 0.2% ropivacaine with 5 mg DEX/ 40 mg MPA
  Arms: Group 1 patients will receive nerve block per standard of care
Procedure: Periarticular Injection (PAI) — Intraoperatively, the surgeon will perform PAI per standard of care with the medications:
  1. 60 ml 0.2% ropivacaine and 10 mg DEX/ 80 mg MPA
  Arms: Group 2 will NOT receive any nerve blocks.
Drug: Ropivacaine — 60 ml 0.2% ropivacaine
Drug: Dex — 10 mg DEX/ 80 mg MPA
  Arms: Group 2 will NOT receive any nerve blocks.

SUMMARY:
This study will assess if preoperative quadratus lumborum block (QLB)/lateral femoral cutaneous nerve block (LFCNB) with ropivacaine and glucocorticoids provide more effective analgesia than periarticular injection (PAI) with the same mixture in total hip arthroplasty (THA).

DETAILED DESCRIPTION:
To support our hypothesis that preoperative quadratus lumborum block (QLB)/lateral femoral cutaneous nerve block (LFCNB) provides more effective analgesia than periarticular injection (PAI) in total hip arthroplasty (THA), we will look at the following outcomes:

Primary outcome: Daily opioid consumption

Secondary outcomes:

Pain intensity and physical functioning while in the hospital: using pain inventory modified from Brief Pain Inventory and Length of hospital stays.

Since both QLB/LFCNB nerve block and PAI techniques are both routinely used as standard of care anesthesia for THA, the study intervention will be the randomization to assign patients to one of these treatment options and assess their response from post-op patient questionnaires and data collection.

When results were entered, the detailed description was updated to reflect the outcome measures used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Elective unilateral primary THA
* All surgical approaches
* American Society of Anesthesiologist (ASA) status I, II and III.

Exclusion Criteria:

* Patient refusal;
* Age less than 18 years
* Those with cognitive dysfunction, psychiatric disorder, or non-English speaking patients that cannot consent or communicate clear understanding of the protocol with research team;
* Coagulopathy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-06-19 (Actual); Study Completion 2021-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinlei Li, MD PhD FASA, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital St Raphael, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group Will NOT Receive Any Nerve Blocks.: Intraoperatively, the surgeon will perform PAI with exactly the same medication as group 1, ie, 60 ml 0.2% ropivacaine and 10 mg DEX/ 80 mg MPA, per standard of care of Surgeon.
  Periarticular Injection (PAI): Intraoperatively, the surgeon will perform PAI per standard of care with the medications:
  1. 60 ml 0.2% ropivacaine and 10 mg DEX/ 80 mg MPA
  Ropivacaine: 60 ml 0.2% ropivacaine
  Dex: 10 mg DEX/ 80 mg MPA
- Group Will Receive Nerve Block Per Standard of Care: Nerve blocks (QLB/LFCNB) to be placed preoperatively with dexamethasone sodium phosphate (DEX) and methylprednisolone acetate (MPA), per standard of care of anesthesia block service.
  1. QLB: 40ml 0.2% ropivacaine with 5 mg DEX/ 40 mg MPA; and
  2. LFCNB: 20ml 0.2% ropivacaine with 5 mg DEX/ 40 mg MPA Preoperatively, Group 1 patients will receive nerve block per standard of care as stated above. Intraoperatively, Group 1 will NOT receive PAI.
  Nerve Block: Nerve blocks (QLB/LFCNB) to be placed preoperatively with DEX/MPA, per standard of care of anesthesia block service.
  1. QLB: 40ml 0.2% ropivacaine with 5 mg DEX/ 40 mg MPA
  2. LFCNB: 20ml 0.2% ropivacaine with 5 mg DEX/ 40 mg MPA
  Ropivacaine: 60 ml 0.2% ropivacaine
Period: Overall Study
Arm/Group | Group Will NOT Receive Any Nerve Blocks. | Group Will Receive Nerve Block Per Standard of Care
Started | 97 | 95
Completed | 95 | 93
Not Completed | 2 | 2
Not completed — immediate postoperative revision | 2 | 2

BASELINE CHARACTERISTICS:
Population: Patients deemed "immediate postoperative revision" were not included in any of the analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Will NOT Receive Any Nerve Blocks. | Group Will Receive Nerve Block Per Standard of Care | Total
Number analyzed (Participants) | 95 | 93 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (10.4) | 61.3 (10.6) | 61.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 44 | 96
  Male | 43 | 49 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 89 | 91 | 180
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 77 | 78 | 155
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 95 | 93 | 188

OUTCOME MEASURES:

1. Primary Outcome: Daily Opioid Consumption
Description: Daily opioid consumption will be monitored during the patient's post surgical hospitalization. Data are presented as milligram morphine equivalent (MME). When the results were entered, the time frame was corrected to reflect the final approved protocol.
Time Frame: Up to 72 hours
Population: Final analysis population (completed from Participant Flow)
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | Group Will NOT Receive Any Nerve Blocks. | Group Will Receive Nerve Block Per Standard of Care
Number analyzed (Participants) | 95 | 93
milligram
  12 hours Post Op | 29.3 (24.0) | 30.8 (22.7)
  24 hours Post Op | 49.6 (36.8) | 51.8 (37.5)
  48 Hours Post Op | 62.1 (47.7) | 67.7 (52.4)
  72 Hours Post Op | 68.6 (58.5) | 71.4 (55.9)
Statistical Analysis 1: Comparison: Group Will NOT Receive Any Nerve Blocks. vs Group Will Receive Nerve Block Per Standard of Care; The primary endpoint was a comparison between groups at 24 hours; Test type: Superiority; p = 0.69, t-test, 2 sided; Mean Difference (Net) = 1.2

2. Secondary Outcome: Change in Pain Intensity While in Hospital
Description: Pain intensity will be assessed using a pain inventory modified from Brief Pain Inventory (BPI). The BPI has a range of 0-10 where: 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-10 = severe pain. Outcome measure was updated at the time of results entry.
Time Frame: Up to 2 days
Population: Final analysis population (completed from Participant Flow)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Will NOT Receive Any Nerve Blocks. | Group Will Receive Nerve Block Per Standard of Care
Number analyzed (Participants) | 95 | 93
units on a scale
  Pre Operation | 4.9 (2.4) | 5.0 (2.1)
  Post Operation Day 1 | 4.2 (2.1) | 4.4 (2.0)
  Post Operation Day 2 | 3.9 (2.3) | 4.0 (1.9)
Statistical Analysis 1: Comparison: Group Will NOT Receive Any Nerve Blocks. vs Group Will Receive Nerve Block Per Standard of Care; Scores were compared at 2 days post operation; Test type: Superiority; p = 0.92, t-test, 2 sided; Mean Difference (Net) = 0.1

3. Secondary Outcome: Length of Stay
Description: The patient's post surgical length of stay in the hospital will be compared between treatment groups. Length of stay is presented as average total hours in hospital.
Time Frame: Up to 5 days
Population: Final analysis population (completed from Participant Flow)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group Will NOT Receive Any Nerve Blocks. | Group Will Receive Nerve Block Per Standard of Care
Number analyzed (Participants) | 95 | 93
hours | 47.2 (24.8) | 46.7 (25.9)
Statistical Analysis 1: Comparison: Group Will NOT Receive Any Nerve Blocks. vs Group Will Receive Nerve Block Per Standard of Care; Test type: Superiority; p = 0.91, t-test, 2 sided; Mean Difference (Net) = 0.5

4. Secondary Outcome: Harris Hip Score
Description: The Harris Hip Score (HHS) assesses post operative conditions following hip surgery. The HHS uses a 100 point score wherethe scores are interpreted as follows: < 70 = poor, 70-79 = fair, 80-89 = good and 90-100 = excellent.
Time Frame: 2 weeks post operation
Population: This measure was not used but the Brief Pain Inventory: Interference scale was used instead.
Arm/Group | Group Will NOT Receive Any Nerve Blocks. | Group Will Receive Nerve Block Per Standard of Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Brief Pain Inventory: Interference
Description: The Brief Pain Inventory: Interference (BPI:I) was used in place of the Harris Hip Score (HHS) to assess post operative conditions following hip surgery. The BPI:I uses a 10 point score where the normal range of scores is: 0 no interference - 10 complete interference.
Time Frame: 2 weeks post operation
Population: Final analysis population (completed from Participant Flow)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Will NOT Receive Any Nerve Blocks. | Group Will Receive Nerve Block Per Standard of Care
Number analyzed (Participants) | 95 | 93
units on a scale
  Pre Operation | 6.2 (2.5) | 6.3 (2.2)
  2 Weeks Post Operation | 2.8 (2.1) | 2.8 (2.1)
Statistical Analysis 1: Comparison: Group Will NOT Receive Any Nerve Blocks. vs Group Will Receive Nerve Block Per Standard of Care; Scores were compared at 2 weeks; Test type: Superiority; p = 0.85, t-test, 2 sided; Mean Difference (Net) = 0.0

ADVERSE EVENTS:
Time Frame: Up to 2 weeks
Arm/Group | Group Will NOT Receive Any Nerve Blocks. | Group Will Receive Nerve Block Per Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/93
Other Adverse Events (participants affected / at risk) | 0/95 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT03977454/Prot_SAP_000.pdf